CLINICAL TRIAL: NCT00668265
Title: A Prospective, Sixteen-Week, Double-Blind, Placebo-Controlled, Trial of Seroquel in Combination With Treatment as Usual in Patients With GAD and Remitted Comorbid Opiate Dependence
Brief Title: Anxiety in Recovering Opiate Dependence
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The study was not completed, the funding sponsor lost interest.
Sponsor: Beth Israel Medical Center (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB # (112-07); IRUSQUET0443
Record Dates: First submitted 2008-04-28; First posted 2008-04-29 (Estimated); Results first posted 2013-02-18 (Estimated); Last update posted 2013-02-18 (Estimated); Status verified 2013-02

CONDITIONS: Generalized Anxiety Disorder; Comorbid Opiate Dependence in Remission; Status Post Methadone-Maintenance Treatment
Keywords: Generalized Anxiety Disorder; Opiate Dependence; Methadone-Maintenance; Drug Addiction Treatment
MeSH Terms: conditions — Generalized Anxiety Disorder; Opioid-Related Disorders | interventions — Quetiapine Fumarate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Seroquel (Experimental)
  Interventions: Drug: Quetiapine

INTERVENTIONS:
Drug: Quetiapine — Dosage is 50 - 300 mg, once daily, at bedtime.
  Other Names: Seroquel

SUMMARY:
This is a 16 week study of the efficacy of quetiapine in treating symptoms of generalized anxiety disorder (GAD) in subjects with comorbid opiate dependence. The study will be conducted in a prospective, randomized, double-blind, and placebo-controlled fashion. Study subjects will be inpatients at a residential drug-treatment facility, enrolled in a 1 year methadone-to-abstinence treatment plan. Subjects will be randomized to receive either quetiapine or placebo in addition to ongoing drug addiction treatment. Subjects will be followed for 16 weeks and a variety of psychometric assessments will be made.

Hypothesis One: Compared to placebo, Quetiapine will demonstrate a greater reduction in symptoms of anxiety in subjects with GAD and remitted comorbid opiate abuse.

Exploratory Hypotheses: Compared to placebo, Quetiapine will demonstrate a greater improvement in psychosocial functioning and compliance with community norms in subjects enrolled in a residential drug addiction treatment facility.

ELIGIBILITY:
Inclusion Criteria:

* Provision of written informed consent
* A diagnosis of opiate dependence as defined by Diagnostic and Statistical Manual of Mental Disorders- Fourth Edition (DSM-IV) during the past two years.
* A diagnosis of generalized anxiety disorder as defined by Diagnostic and Statistical Manual of Mental Disorders- Fourth Edition (DSM-IV) within the past 6 months.
* Males and females aged 21-55 years
* Female patients of childbearing potential must be using a reliable method of contraception and have a negative urine human chorionic gonadotropin (HCG) test at enrollment
* Able to understand and comply with the requirements of the study
* Subjects must be free of illicit drug use for the past 3 months
* Subjects must have received methadone maintenance therapy for at least 3 months, and have been at least 2 weeks methadone-free
* Good health, as assessed by medical history, physical examination and laboratory tests

Exclusion Criteria:

* Pregnancy or lactation
* Current diagnosis of any Axis I disorder other than GAD, substance dependence in remission, or nicotine dependence
* Patients who, in the opinion of the investigator, pose an imminent risk of suicide or a danger to self or others
* Known intolerance or lack of response to quetiapine fumarate, as judged by the investigator
* Use of any of the following cytochrome P450 3A4 inhibitors in the 14 days preceding enrolment including but not limited to: ketoconazole, itraconazole, fluconazole, erythromycin, clarithromycin, troleandomycin, indinavir, nelfinavir, ritonavir, fluvoxamine and saquinavir
* Use of any of the following cytochrome P450 inducers in the 14 days preceding enrollment including but not limited to: phenytoin, carbamazepine, barbiturates, rifampin, St. John's Wort, and glucocorticoids
* Administration of a depot antipsychotic injection within one dosing interval (for the depot) before randomisation
* Medical conditions that would affect absorption, distribution, metabolism, or excretion of study treatment
* Unstable or inadequately treated medical illness (e.g. diabetes, angina pectoris, hypertension) as judged by the investigator
* Involvement in the planning and conduct of the study
* Previous enrollment or randomisation of treatment in the present study.
* Participation in another drug trial within 4 weeks prior enrollment into this study or longer in accordance with local requirements
* A patient with Diabetes Mellitus (DM) fulfilling one of the following criteria:
* Unstable DM defined as enrollment glycosylated hemoglobin (HbA1c) >8.5%.
* Admitted to hospital for treatment of DM or DM related illness in past 12 weeks.
* Not under physician care for DM
* Physician responsible for patient's DM care has not indicated that patient's DM is controlled.
* Physician responsible for patient's DM care has not approved patient's participation in the study
* Has not been on the same dose of oral hypoglycaemic drug(s) and/or diet for the 4 weeks prior to randomization. For thiazolidinediones (glitazones) this period should not be less than 8 weeks.
* Taking insulin whose daily dose on one occasion in the past 4 weeks has been more than 10% above or below their mean dose in the preceding 4 weeks Note: If a diabetic patient meets one of these criteria, the patient is to be excluded even if the treating physician believes that the patient is stable and can participate in the study.
* An absolute neutrophil count (ANC) of 1.5 x 109 per liter
* Positive urine drug screening test for drugs of abuse

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2008-01; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sean Chappin, M.D., Principal Investigator — Beth Israel Medical Center
Locations (1):
- Su Casa Methadone-to-Abstinence Rehabilitation, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was initiated in 2007 adn terminated in 2010 due to PI's departure. All recrutiement took place at Su Casa residential treatment facility in New York City. All recruitment was done by the PI.
Pre-assignment Details: The subjects were individuals with opiate addiction on agonist therapy. After recruitement subjects underwent methadone taper as inpatients. Most subjects left the study because they signed out of the Su Casa Program and did not complete their methadone taper.
Groups:
- Quetiapine Arm: The participants were scheduled to receive Quetiapine, initially at a dose of 50 mg qHS for 2 days, followed by 100 mg qHS for 2 days, and then raised to a target dose of 150 mg qHS. Patients who do not tolerate that dose were titrated downwards in 50 mg increments until a tolerable dose is achieved. Medication dosage was further adjusted as necessary during the course of the study.
  Concomitant Medications:
  Concomitant psychotropic medications were not allowed. Concomitant medications for treatment of physical illnesses other than those indicated in the Exclusion Criteria were allowed
- Placebo Arm: The subjects in the placebo arm received inactive pills in identical blister packs
Period: Overall Study
Arm/Group | Quetiapine Arm | Placebo Arm
Started | 9 | 5
Completed | 0 (The PI left, no records avaialable; the number of subjects who completed the study is not known) | 0 (The PI left, no records avaialable; the number of subjects who completed the study is not known)
Not Completed | 9 | 5

BASELINE CHARACTERISTICS:
Groups:
- Quetiapine: Subjects on MMTP receiving quetiapine
- Placebo: Subjects on methadone maintenance receiving placebo while inpatients in a methadone treatment facility Su Casa
- Total: Total of all reporting groups
Arm/Group | Quetiapine | Placebo | Total
Number analyzed (Participants) | 9 | 5 | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 9 | 5 | 14
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 43 (7.0) | 45 (9) | 43.8 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 7 | 4 | 11
Region of Enrollment [Number; unit: participants]
  United States | 9 | 5 | 14

OUTCOME MEASURES:

1. Primary Outcome: Hamilton Anxiety Scale at 16 Weeks
Description: Hamilton anxiety scale -- a well known quantitative measure for assessment of anxiety
Time Frame: 16 weeks
Population: Data was not analyzed: PI left the institution and the study was terminated
Arm/Group | Quetiapine | Placebo
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Beck Depression Inventory at 16 Weeks
Description: To compare the effect of Quetiapine vs. placebo on symptoms of negative mood in patients with GAD and comorbid opiate abuse in remission.
Time Frame: 16 weeks
Population: Data were not analyzed. PI left institution, and did not respond to attempts top contact him.
Arm/Group | Quetiapine Arm | Placebo Arm
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Description: Adverse events are not available. PI left the institution and did not respond to attempts to contact him.
Groups:
- Quetiapine: Active treatment arm for subjects on MMTP in Su Casa residence
- Placebo: Placebo arm for subjects on MMTP in Su Casa Residence
Arm/Group | Quetiapine | Placebo
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes